CLINICAL TRIAL: NCT02621151
Title: A Phase II Trial of MK3475 in Combination With Gemcitabine and Concurrent Hypofractionated Radiation Therapy as Bladder Sparing Treatment for Muscle-Invasive Urothelial Cancer of the Bladder
Brief Title: Pembrolizumab (MK3475), Gemcitabine, and Concurrent Hypofractionated Radiation Therapy for Muscle-Invasive Urothelial Cancer of the Bladder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00220
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Muscle-invasive Urothelial Cancer of the Bladder
Keywords: combination therapy; immunotherapy; immune checkpoint inhibition
MeSH Terms: interventions — pembrolizumab; Transurethral Resection of Bladder; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab, Gemcitabine, and RT (Experimental): * Lead-in single dose Pembrolizumab 200 mg, intravenously (IV)
  * Transurethral Resection of Bladder Tumor (TURBT) at pre-RT (maximal) and completion of therapy (diagnostic)
  * External Beam Radiation Therapy (EBRT) - 52 Gy in 20 fractions over 4 weeks (1 fraction = 2.6 Gy)
  * Gemcitabine 27 mg/m^2 IV twice weekly for 4 weeks concurrent with EBRT
  * Pembrolizumab 200 mg IV every 3 weeks for total 3 doses starting day 1 of EBRT
  Interventions: Biological: Pembrolizumab; Procedure: Transurethral Resection of Bladder Tumor; Drug: Gemcitabine; Radiation: External Beam Radiation Therapy

INTERVENTIONS:
Biological: Pembrolizumab
  Other Names: MK3475; Keytruda
Procedure: Transurethral Resection of Bladder Tumor
Drug: Gemcitabine
  Other Names: Gemzar
Radiation: External Beam Radiation Therapy

SUMMARY:
This trial is to assess the efficacy of pembrolizumab (MK3475) added to concurrent radiation and gemcitabine in the management of patients with muscle-invasive urothelial cancer who are not candidates for or decline radical cystectomy.

DETAILED DESCRIPTION:
The investigators hypothesize that the addition of immune checkpoint inhibition with pembrolizumab, an anti-PD-1 inhibitor, to chemo-radiation therapy to the bladder may work to both increase eradication of local tumor as well as distant micrometastases through heightened immune surveillance.

Due to the lack of a previous phase I trial establishing the safety of this combination (pembrolizumab, gemcitabine, and radiation therapy (RT)), an initial safety lead-in cohort of 3 to 6 patients is enrolled for assessing dose-limiting toxicities. Similar to the Phase I 3+3 design, if there is no or only one patient in that cohort experiencing a dose-limiting toxicity, the trial continues to the Phase II part to enroll additional 48 patients for efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed muscle-invasive urothelial cancer of the bladder within 60 days of study enrollment. Patients must be willing to provide a TURBT specimen during screening and prior to enrollment if adequate specimen (FFPE tissue block or 20 unstained slides) from initial TURBT documenting muscle-invasive urothelial bladder cancer is not available.
* Clinical stage T2-T4a, N0, M0 urothelial bladder cancer.
* Deemed to not be a candidate for radical cystectomy by attending urologic oncologist or refuse radical cystectomy.
* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group Performance Scale.
* Demonstrate adequate organ function as defined below, all screening labs should be performed within 10 days of protocol enrollment.

  * Absolute neutrophil count >= 1,500 /mcL;
  * Platelets >= 100,000 /mcL;
  * Hemoglobin >= 9.0 g/dL;
  * Serum creatinine <=1.5 x upper limit of normal (ULN) or calculated creatinine clearance >= 30 mL/min as calculated by Cockcrof-Gault formaulae or by 24 hour urine collection;
  * Serum total bilirubin <=1.5 x ULN or direct bilirubin <= ULN for subjects with total bilirubin levels > 1.5 x ULN;
  * Aspartate aminotransferase and alanine aminotransferase <= 1.5 x ULN;
  * Albumin >= 2.5 mg/dL;
  * International normalized ratio or prothrombin time (PT) <= 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial prothrombin time (PTT) is within therapeutic range of intended use of anticoagulants;
  * Activated Partial Thromboplastin Time (aPTT) <= 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Has received prior targeted small molecule therapy, radiation therapy or systemic chemotherapy for urothelial bladder cancer including neoadjuvant chemotherapy. Prior intravesical chemotherapy or intravesical immunotherapy is permissible, however, no prior intravesical therapy is permitted within 4 weeks of study enrollment; adjuvant therapy is not permitted.
* Has received prior pelvic radiation therapy.
* Has a history of inflammatory bowel disease or history of scleroderma.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Any prior history of invasive malignancy within the past 5 years except non-melanoma skin cancer, carcinoma in-situ, localized prostate cancer without biochemical recurrence following definitive treatment.
* Has any history of inflammatory bowel disease or scleroderma.
* Has other active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of Guillain-Barre Syndrome or Stevens-Johnson Syndrome
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Minas Economides, MD, Principal Investigator — NYU Langone Health
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - NYU Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: [contact information for PI or designee]. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to minas.economides@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab, Gemcitabine, and RT: * Lead-in single dose Pembrolizumab 200 mg, intravenously (IV)
  * Transurethral Resection of Bladder Tumor (TURBT) at pre-RT (maximal) and completion of therapy (diagnostic)
  * External Beam Radiation Therapy (EBRT) - 52 Gy in 20 fractions over 4 weeks (1 fraction = 2.6 Gy)
  * Gemcitabine 27 mg/m^2 IV twice weekly for 4 weeks concurrent with EBRT
  * Pembrolizumab 200 mg IV every 3 weeks for total 3 doses starting day 1 of EBRT
  Pembrolizumab
  Transurethral Resection of Bladder Tumor
  Gemcitabine
  External Beam Radiation Therapy
Period: Overall Study
Arm/Group | Pembrolizumab, Gemcitabine, and RT
Started | 60
Completed | 54
Not Completed | 6
Not completed — Not eligible for trial | 6

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab, Gemcitabine, and RT
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 73.6 [51.2 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 45
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Two-year Bladder-intact Disease-free Survival
Description: Bladder-intact disease-free survival is defined as the time from initiation of protocol therapy until the first occurrence of muscle-invasive bladder cancer recurrence, regional pelvic recurrence, distant metastases, bladder cancer-related death, or cystectomy.
Time Frame: 2 years
Population: The analysis focused on the efficacy cohort and did not include the safety lead-in cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab, Gemcitabine, and RT
Number analyzed (Participants) | 48
percentage of participants | 60 [45 to 73]

2. Secondary Outcome: Complete Response (CR) Rate
Description: The CR rate is the percentage of patients who have achieved CR. At the completion of protocol therapy, patients undergo standard cystoscopy, exam under anesthesia and transurethral resection of bladder tumor to document pathologic response. CR requires no tumor palpable on bimanual examination under anesthesia, no tumor visible on cystoscopy, negative tumor site biopsy, and negative urine cytology.
Time Frame: up to 21 weeks
Population: The analysis focused on the efficacy cohort and did not include the safety lead-in cohort.
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab, Gemcitabine, and RT
Number analyzed (Participants) | 48
percentage of participants | 56

3. Secondary Outcome: Percentage of Participants Who Survived at Study Completion
Time Frame: up to 5 years
Population: The analysis focused on the efficacy cohort and did not include the safety lead-in cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab, Gemcitabine, and RT
Number analyzed (Participants) | 48
percentage of participants | 83 [68.9 to 91.1]

4. Secondary Outcome: Percentage of Participants Who Achieved Metastasis-free Survival at Study Completion
Description: Metastasis-free survival is defined as not having developed radiographic distant metastases.
Time Frame: up to 5 years
Population: The analysis focused on the efficacy cohort and did not include the safety lead-in cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab, Gemcitabine, and RT
Number analyzed (Participants) | 48
percentage of participants | 84 [70 to 92]

ADVERSE EVENTS:
Time Frame: AEs and SAEs assessed for 16 weeks (consent through 30 days post treatment); All cause mortality assessed throughout the 5 year study period
Description: investigator assessment at each treatment and follow-up visit
Arm/Group | Pembrolizumab, Gemcitabine, and RT
All-Cause Mortality (participants affected / at risk) | 16/54
Serious Adverse Events (participants affected / at risk) | 15/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab, Gemcitabine, and RT (N=54)
Abdominal Pain (Gastrointestinal disorders) | 13
Aspartate Aminotransferase Increased (Investigations) | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Chest Pain (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Colonic Perforation (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Protein Losing Enteropathy (Gastrointestinal disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 6
Immune System Disorders - Other (Immune system disorders) | 1
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 3
Urinary Tract Infection (Renal and urinary disorders) | 13
Urinary Tract Obstruction (Renal and urinary disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab, Gemcitabine, and RT (N=54)
Abdominal Distention (Gastrointestinal disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Alanine Aminotransferace Increased (Investigations) | 9
Anemia (Blood and lymphatic system disorders) | 18
Anorexia (Metabolism and nutrition disorders) | 15
Anxiety (Psychiatric disorders) | 1
Arthalgia (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 9
Bladder Spasm (Renal and urinary disorders) | 11
Bloating (Gastrointestinal disorders) | 3
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1
Blood Bilirubin Increased (Investigations) | 1
Bronchial Infection (Respiratory, thoracic and mediastinal disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Cardiac Disorders - Other (Cardiac disorders) | 1
Chills (General disorders) | 5
Chronic Kidney Disease (Renal and urinary disorders) | 1
Cold (General disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Creatinine Increase (Investigations) | 6
Cystitis Noninfective (Renal and urinary disorders) | 1
Delirium (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 25
Dizziness (Nervous system disorders) | 7
Dry Mouth (Gastrointestinal disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Dysuria (Renal and urinary disorders) | 2
Otitis Media (Ear and labyrinth disorders) | 1
Ear And Labyrinth Disorders - Other (Ear and labyrinth disorders) | 1
Elevated Lft (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 31
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Fecal Incontinence (Gastrointestinal disorders) | 1
Fever (General disorders) | 8
Flatulence (Gastrointestinal disorders) | 4
Flu Like Symptoms (General disorders) | 2
Gait Disturbance (General disorders) | 2
Gas (Gastrointestinal disorders) | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 10
General Disorders And Administration Site Conditions - Other (General disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4
Fecal Urgency (Gastrointestinal disorders) | 2
Diverticulosis (Gastrointestinal disorders) | 1
Loose Stool (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 7
Hematuria (Renal and urinary disorders) | 17
Hemorrhoids (Gastrointestinal disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypertension (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Cardiac disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Kidney Infection (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 2
Insomnia (Psychiatric disorders) | 2
Intraoperative Urinary Injury (Injury, poisoning and procedural complications) | 1
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 1
Irritability (General disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Lower Abdominal Discomfort (Gastrointestinal disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 3
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 4
Malaise (General disorders) | 2
Metabolism And Nutrition Disorders, Other (Metabolism and nutrition disorders) | 1
Musocal Infection (Infections and infestations) | 1
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 27
Neutropenia (Blood and lymphatic system disorders) | 8
Pain (General disorders) | 8
Paresthesia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Pharyngitis (Infections and infestations) | 1
Platelet Count Decreased (Investigations) | 16
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Proctitis (Gastrointestinal disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14
Rectal Mucus Discharge (Gastrointestinal disorders) | 1
Rectal Pain (Gastrointestinal disorders) | 3
Rectal Spasms (Gastrointestinal disorders) | 1
Rectal Ulcer (Gastrointestinal disorders) | 1
Rectal Urgency (Gastrointestinal disorders) | 1
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 6
Retinopathy (Eye disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 2
Sinus Tachycardia (Cardiac disorders) | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Skin And Other Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 3
Skin Infection (Skin and subcutaneous tissue disorders) | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2
Stomach Pain (Gastrointestinal disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 1
Thromboembolitic Event (Vascular disorders) | 1
Tooth Infection (Infections and infestations) | 1
Urinary Frequency (Renal and urinary disorders) | 21
Urinary Incontinence (Renal and urinary disorders) | 8
Urinary Retention (Renal and urinary disorders) | 4
Urinary Tract Pain (Renal and urinary disorders) | 19
Urinary Urgency (Renal and urinary disorders) | 8
Vascular Disorder, Other (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Weight Gain (Investigations) | 1
White Blood Cell Decreased (Blood and lymphatic system disorders) | 8
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT02621151/Prot_SAP_000.pdf